CLINICAL TRIAL: NCT02292420
Title: The Normal Reference Values of Pulse Oximetry Plethymographic Waveform Parameters
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jun Xu, Emergency Department, Peking Union Medical College Hospital
Other Study IDs: S-743
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Pulse Oximetry Plethymographic Waveform; Area Under Curve; Amplitude
Keywords: pulse oximetry plethymographic waveform; area under curve; amplitude

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the normal reference values of pulse oximetry plethymographic waveform parameters in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

Healty adults; Comply with ethical requirements and signed informed consent.

Exclusion Criteria:

Leuconychia; Stained fingernails; Diseases that have an impact on the blood flow of the peripheral tissue (such as Raynaud's phenomenon, vasculitis and so on); Any conditions the study physicians believe not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 1019 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
parameters of pulse oximetry plethymographic waveform | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Xuezhong Yu, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China